CLINICAL TRIAL: NCT02665650
Title: A Phase 1b Dose Escalation Study to Assess the Safety of AFM13 in Combination With Pembrolizumab in Patients With Relapsed or Refractory Classical Hodgkin Lymphoma (KEYNOTE- 206)
Brief Title: Study of the Combination of AFM13 and Pembrolizumab in Patients With Relapsed or Refractory Classical Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affimed GmbH (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFM13-103
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-01

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — AFM13; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AFM13 + Pembrolizumab (Experimental): Participants receive AFM13 in escalating doses intravenously (IV) for up to 25 weeks, pembrolizumab as a fixed dose intravenously (IV) for up to 52 weeks.
  Interventions: Biological: AFM13; Biological: Pembrolizumab

INTERVENTIONS:
Biological: AFM13
Biological: Pembrolizumab
  Other Names: MK-3475; Keytruda

SUMMARY:
The purpose of this study is to establish a dosing regimen for the combination therapy of AFM13 and pembrolizumab (MK-3475) in patients with relapsed or refractory (R/R) Hodgkin Lymphoma (HL) and to assess the safety and tolerability of this combination therapy.

ELIGIBILITY:
Main Inclusion Criteria:

1. Diagnosis of CD30+ classical Hodgkin lymphoma reconfirmed by histopathology. Note: where reconfirmation is not possible, patients will still be eligible where they have confirmation clearly documented in their medical records.
2. Relapsed or refractory disease after standard therapy including brentuximab vedotin (Adcetris®).
3. Completion of, if applicable, radiotherapy, chemotherapy, antibodies and immunoconjugates including brentuximab vedotin and/or another investigational drug which could interact with this trial not less than 4 weeks (or 5 half-lives of the drug, whichever occurs later) prior to first dose of study drug. Cessation of small molecule tyrosine kinase inhibitors must be at least 7 days prior to first dose of study drug.
4. Completion of, if applicable, an autologous stem cell transplantation (ASCT) at least 3 months prior to first dose of study drug.
5. Eastern Cooperative Oncology Group (ECOG) performance score (PS) <2.

Main Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or if the patient has previously participated in MK-3475 clinical trials.
3. Has received a live-virus vaccination within 30 days of planned treatment start. Note: Seasonal flu vaccines that do not contain live virus are permitted.
4. Prior allogeneic stem cell transplantation (SCT) within the last 5 years.
5. Major surgery within 4 weeks prior to first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2019-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing dose limiting toxicity (DLT) during combination treatment | Up to 9 months

SECONDARY OUTCOMES:
Number and frequency of adverse events | Up to 30 months
Objective response rate (ORR) | Up to 30 months

CONTACTS AND LOCATIONS:
Locations (18):
- United States (14):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - University of Miami Sylvester Comprehensive Cancer Center, Coral Gables, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Medical Center, St Louis, Missouri
  - Providence Portland Medical Center, Providence Cancer Center, Portland, Oregon
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Spain (4):
  - Institut Catala d'Oncologia (ICO) L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Fundacion Privada Instituto de Investigacion Oncologica de Vall Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Servicio de Hematologia, Madrid
  - Salamanca University Hospital, Salamanca

REFERENCES:
- [Derived] Bartlett NL, Herrera AF, Domingo-Domenech E, Mehta A, Forero-Torres A, Garcia-Sanz R, Armand P, Devata S, Izquierdo AR, Lossos IS, Reeder C, Sher T, Chen R, Schwarz SE, Alland L, Strassz A, Prier K, Choe-Juliak C, Ansell SM. A phase 1b study of AFM13 in combination with pembrolizumab in patients with relapsed or refractory Hodgkin lymphoma. Blood. 2020 Nov 19;136(21):2401-2409. doi: 10.1182/blood.2019004701. PMID 32730586